CLINICAL TRIAL: NCT05692414
Title: Preoperative Carbohydrate Loading in Bariatric Surgery - Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Andrii Bilyk, Student, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKBBN/200/2020
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Bariatric Surgery; Carbohydrate Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative carbohydrate loaded patients (Experimental)
  Interventions: Dietary Supplement: Preoperative carbohydrate drink
- Conventional fasting protocol (No Intervention)

INTERVENTIONS:
Dietary Supplement: Preoperative carbohydrate drink — Allocation will be performed using an alternating weeks scheme. Patients undergoing surgery in the first week will be included in the control group and follow a conventional fasting protocol. However, patients undergoing surgery the following week will be included in the intervention group and take 800 ml of CHO drink on the day before surgery and 400 ml on the surgery day no later than 6 hours before the procedure.
  Arms: Preoperative carbohydrate loaded patients

SUMMARY:
Insulin resistance is a key feature of postoperative metabolism, leading to decreased glucose absorption in adipose tissue and skeletal muscle, with an increased glucose release due to hepatic gluconeogenesis and hyperglycemia. Development of insulin resistance is associated with increased length of hospital stay (LOS), morbidity, and mortality. One of the strategies employed to reduce the postoperative stress response and perioperative insulin resistance includes the reduction of the preoperative fasting time via preoperative carbohydrate oral (CHO) drink. Preoperative carbohydrate intake is an integral part of the Enhanced Recovery After Surgery (ERAS) protocol and previous studies have shown that preoperative carbohydrate loading can increase patient comfort. Although ERAS protocols are increasingly used and implemented in bariatric surgery centres specific components of these protocols, such as preoperative oral carbohydrate nutrition, have not yet been rigorously analyzed.

The aim of this prospective study is to compare the differences in patient outcomes between preoperative CHO loading and a conventional fasting protocol. The secondary aim is to perform a subgroup analysis of Roux-en-Y bypass and sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo surgery at the Elective Surgery Clinic of the University Clinical Centre in Gdansk, Poland.

Exclusion Criteria:

* Patients who will be unable or will refuse to express informed concern

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Glucose level | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Centre in Gdansk, Gdansk, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: Undecided